CLINICAL TRIAL: NCT06400524
Title: Assessment of Myocardial Function, (Peripheral) Endothelial Function and Perfusion in Early and Advanced Disease Stages of Hypertrophic Cardiomyopathy
Brief Title: Assessment of Cardiac Function, Microvascular Function and Cardiac Perfusion in Different Disease Stages of Hypertrophic Cardiomyopathy
Acronym: FUSION-HCM
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Tjeerd Germans, Dr., Amsterdam UMC, location VUmc
Other Study IDs: NL83573.018.23
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Hypertrophic Cardiomyopathy; Hypertrophic Cardiomyopathy, Obstructive
Keywords: hypertrophic cardiomyopathy; perfusion; endothelial function
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy controls
- Mutation carriers
- Mild hypertrophy
- Overt hypertrophy

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a genetic disorder characterized by asymmetric hypertrophy of the heart in absence of loading conditions like hypertension. The genetic mutation underlying HCM sets in motion a cascade of functional and metabolic changes ultimately leading to disease. HCM patients often have microvascular dysfunction and myocardial perfusion deficits, of which the aetiology has not been elucidated. Whether these changes are secondary to remodelling or primarily caused by endothelial dysfunction is unclear. As the pathomechanism of HCM is thought to be a cascade of changes, it is important to gain more insight in the perfusion and endothelial function changes throughout different stages of disease: no phenotype, mild phenotype, and advanced HCM phenotype. In this study we aim to investigate these changes in the two most common genetic mutations.

ELIGIBILITY:
Inclusion Criteria:

One of below:

* MYBPC3 mutation carrier
* MYH7 mutation carrier
* Genotype-negative first degree relative of a MYBPC3 or MYH7 mutation carrier

All of the following criteria:

* For the mutation carrier group: ≥18 years old
* For the genotype-negative group: ≥30 years old

MYBPC3 and MYH7 mutation carriers will be designated to one of three groups based on their maximum wall thickness, measured by echocardiography and MRI:

* No phenotype: MWT <12mm
* Mild Phenotype: MWT ≥12 until <15mm
* HCM phenotype: MWT ≥15mm

Exclusion Criteria:

* ≥70 years old
* Insulin-dependent diabetes mellitus
* Pregnancy
* Smoking
* Claustrophobia
* Pacemaker/ICD
* Renal insufficiency <30 GFR
* Hypertension (systolic >140mmHg or diastolic >90mmHg)
* For the genotype negative group, no phenotype group, and mild phenotype group: the use of blood pressure medication (diuretics, beta-blockers, ACE-inhibitors, angiotensin II receptor blockers, calcium channel blockers, alpha blockers)
* For the HCM phenotype group: when it is unsafe to withhold from blood pressure medication (as specified above) for two days, as assessed by their own cardiologist
* Left ventricular outflow tract gradient > 50mmHg
* Aortic valve disease
* Left bundle branch block
* (History of) Obstructive coronary artery disease
* Chronic atrial fibrillation
* Hormone replacement therapy
* Second or third-degree AV-block, sick-sinussyndrome, prolonged QT-interval
* Asthma and other obstructive pulmonary diseases
* Previous adverse reaction to adenosine or dotarem

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Potential study subjects are recruited from different hospitals and will be invited to the VUmc. Our research consortium consists of cardiologists and cardiogeneticists who will spread our call for participants to their patients. We will also work together with the HCM patient organization. Potential study subjects will be invited to contact us by phone or e-mail, after which an information letter will be sent. If someone is interested in participation in the study, they will be invited to the VUmc to sign informed consent and undergo day 1 of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
myocardial blood flow | 1 month
  assessed by PET and CMR
peripheral endothelial function | 1 month
  assessed by EndoPAT and LASCA

SECONDARY OUTCOMES:
Tissue characterization | 1 month
  assessed by CMR
Diastolic dysfunction | 1 month
  assessed by echocardiography
Fibrosis | 1 month
  assessed by CMR

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC - location VUmc, Amsterdam, North Holland, Netherlands